CLINICAL TRIAL: NCT01597089
Title: Detection of Respiratory Viruses in Upper and Lower Respiratory Tract Specimens Using a Rapid Multiplex PCR
Brief Title: Detecting Respiratory Viruses in Upper and Lower Respiratory Tract Samples
Status: Terminated | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 120125; 12-CC-0125
Record Dates: First submitted 2012-05-10; First posted 2012-05-11 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05-01

CONDITIONS: Respiratory Viruses
Keywords: Specificity; Bronchoalveolar Lavage; Film Array Assay; Nasopharyngeal Swab; Sensitivity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Background:

- Bronchoalveolar lavage (BAL) is a procedure where a tube is passed through the mouth or nose into the lungs. Fluid is squirted through the tube into a part of the lung and then collected for examination. It is used to detect respiratory viruses. BAL is a relatively invasive procedure, and researchers want to test the accuracy of other procedures that do not involve collecting fluid from the lungs. The nasopharynx is the area of the upper throat that lies behind the nose. Researchers want to see if a swab taken from this area is as accurate as a BAL sample.

Objectives:

- To see if a nasopharynx swab can be used to detect respiratory viruses as well as BAL samples.

Eligibility:

- Individuals at least 12 years of age who will have a bronchoscopy to collect a BAL sample to test for respiratory viruses.

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will have a BAL sample collected.
* Participants will then have a nasopharynx swab. The swab will be inserted into the nose, left in place for up to 10 seconds, and then removed

DETAILED DESCRIPTION:
Bronchoalveolar lavage (BAL) specimens can be used for the detection of respiratory viruses. Although bronchoscopy is relatively safe, it still has inherent risks to the subject. Nasopharyngeal (NP) swab specimens are easy to collect and are minimally invasive for the subject. We will use a rapid multiplex polymerase chain reaction (PCR) to detect respiratory viruses in paired BAL and NP specimens to determine if either specimen is more likely to be positive. The study population will include all patients undergoing bronchoscopy for clinical indications at the Clinical Center. This is a prospective observational study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 12 years or above
* Scheduled for clinically indicated bronchoscopy for the collection of a BAL specimen and will have respiratory virus PCR ordered on the BAL specimen as part of their ongoing care at the NIH Clinical Center.
* Must agree to allow the storage of their samples (BAL and NP) for use in future research.

EXCLUSION CRITERIA:

None

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-09-01; Study Completion 2018-05-01

PRIMARY OUTCOMES:
The presence or absence of one or more of the 15 respiratory viruses in upper or lower respiratory tract samples using the FilmArray assay. | Within 30 days after collection

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Chertow, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kuypers J, Campbell AP, Cent A, Corey L, Boeckh M. Comparison of conventional and molecular detection of respiratory viruses in hematopoietic cell transplant recipients. Transpl Infect Dis. 2009 Aug;11(4):298-303. doi: 10.1111/j.1399-3062.2009.00400.x. Epub 2009 May 11. PMID 19453994
- [Background] Blyth CC, Iredell JR, Dwyer DE. Rapid-test sensitivity for novel swine-origin influenza A (H1N1) virus in humans. N Engl J Med. 2009 Dec 17;361(25):2493. doi: 10.1056/NEJMc0909049. Epub 2009 Nov 18. No abstract available. PMID 19923563
- [Background] Soccal PM, Aubert JD, Bridevaux PO, Garbino J, Thomas Y, Rochat T, Rochat TS, Meylan P, Tapparel C, Kaiser L. Upper and lower respiratory tract viral infections and acute graft rejection in lung transplant recipients. Clin Infect Dis. 2010 Jul 15;51(2):163-70. doi: 10.1086/653529. PMID 20524853